CLINICAL TRIAL: NCT02675491
Title: Phase 1 Study of DS-6051b in Japanese Subjects With Advanced Solid Malignant Tumors Harboring Either a ROS1 or NTRK Fusion Gene
Brief Title: Phase 1 Study of DS-6051b in Japanese Subjects With Advanced Solid Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS6051-A-J102; 153111 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Malignant Tumors
Keywords: Advanced solid tumor; DS-6051b; ROS1; NTRK; refractory to standard therapy; no standard therapy

ARMS (1):
- DS-6051b (Experimental): Drug: DS-6051b 400 mg or 800 mg daily
  Interventions: Drug: DS-6051b

INTERVENTIONS:
Drug: DS-6051b — Drug: DS-6051b 400 mg or 800 mg daily

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, and pharmacokinetics of DS-6051b in Japanese subjects with advanced solid malignant tumors harboring either a ROS1 or NTRK fusion gene.

DETAILED DESCRIPTION:
This study is single arm study with DS-6051b in approximately 9 subjects with advanced solid malignant tumors harboring either a ROS1 or NTRK fusion gene. Safety and tolerability, pharmacokinetics (PK), maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) and preliminary efficacy of DS-6051b will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid malignant tumors that are refractory to standard therapy or for which no standard therapy is available.
* An Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.

Exclusion Criteria:

* Previously had or currently has any of the following diseases:

Cardiac failure (NYHA Functional Classification ≥ Class III), myocardial infarction, cerebral infarction, unstable angina, arrhythmia requiring treatment, coronary/peripheral artery disease, pulmonary thrombosis, uncontrolled deep vein thrombosis, clinically severe thromboembolic event, or autoimmune disease requiring treatment.

* Previously had or currently has clinically severe pulmonary disease (eg, interstitial pneumonia, pneumonitis, pulmonary fibrosis, radiation pneumonia).
* Severe or uncontrolled concomitant disease.
* Clinically active brain metastases or central nervous system tumor requiring steroid or anticonvulsant treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
number and severity of adverse events | Day 1 through 28 days after last dose
  number and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
Cmax of DS-6051a | Days 1 and 15 of Cycle 1
  Maximum concentration (Cmax), time to maximum plasma concentration (Tmax), area under the concentration-time curve (AUC) and CL/F for DS-6051a (a free base form of DS-6051b) will be assessed on Days 1 and 15 of Cycle 1.
Tmax of DS-6051a | Days 1 and 15 of Cycle 1
  Maximum concentration (Cmax), time to maximum plasma concentration (Tmax), area under the concentration-time curve (AUC) and CL/F for DS-6051a (a free base form of DS-6051b) will be assessed on Days 1 and 15 of Cycle 1.
AUC of DS-6051a | Days 1 and 15 of Cycle 1
  Maximum concentration (Cmax), time to maximum plasma concentration (Tmax), area under the concentration-time curve (AUC) and CL/F for DS-6051a (a free base form of DS-6051b) will be assessed on Days 1 and 15 of Cycle 1.
clearance (CL/F) of DS-6051a | Days 1 and 15 of Cycle 1
  Maximum concentration (Cmax), time to maximum plasma concentration (Tmax), area under the concentration-time curve (AUC) and CL/F for DS-6051a (a free base form of DS-6051b) will be assessed on Days 1 and 15 of Cycle 1.
Number of participants with dose-limiting toxicities | 21 days following the first dose of treatment
  to determine maximum tolerated dose/recommended phase 2 dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (3):
- Japan (3):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kinki University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/